CLINICAL TRIAL: NCT05277285
Title: Hydrogen Sulfate Guided Therapy With STS for COVID-19 Patients in Need of Critical Care: The H4COVID Open-label, Randomized, Triple-arm Trial
Brief Title: STS Administration on Coronavirus Disease (COVID-19) Patients in Critical Care
Acronym: H4COVID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H4COVID
Record Dates: First submitted 2022-03-10; First posted 2022-03-14 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Virus Diseases; Corona Virus Infection
Keywords: COVID-19; SARS-CoV-2; Hydrogen Sulfide; Sodium Thiosulfate; Hydrogen Sulfide donor
MeSH Terms: conditions — COVID-19; Virus Diseases; Coronavirus Infections | interventions — sodium thiosulfate; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Treatment (No Intervention): The standard treatment includes the application of mechanical ventilation and / or support with the administration of inotropes and / or extracorporeal oxygenation (ECMO) and the intravenous administration of fluids and dexamethasone. The administration of any other immunosuppressive therapy, including tocilizumab and / or antimicrobials at the discretion of the therapists, is permitted.
- One intravenous 12.5 gr STS - Treatment Group 1 (Experimental): Patients will receive standard treatment and one intravenous (iv)12.5 gr STS in 60 minutes continuous intravenous infusion. STS is dissolved in a final volume of 100ml N/S 0.9% w/v,
  Interventions: Drug: Sodium Thiosulfate 25% Solution for Injection
- Three intravenous doses of 12.5 gr STS - Treatment Group 2 (Experimental): Patients will receive standard treatment and three intravenous doses of 12.5 g STS. STS is dissolved in a final volume of 100ml N/S 0.9% w/v. Each dose will be given in 60 minutes of continuous intravenous infusion with 48 hours intervals between each dose.
  Interventions: Drug: Sodium Thiosulfate 25% Solution for Injection

INTERVENTIONS:
Drug: Sodium Thiosulfate 25% Solution for Injection — The drug will be administered via continuous infusion after being diluted to a concentration 12.5 gr/100ml
  Other Names: NATRIUMTHIOSULFAT 25%
  Arms: One intravenous 12.5 gr STS - Treatment Group 1; Three intravenous doses of 12.5 gr STS - Treatment Group 2

SUMMARY:
The primary purpose is to describe the safety of administration of three doses of STS to critically ill patients with confirmed COVID-19. A secondary purpose is to describe data on the clinical efficacy of administration of up to three doses of STS in critically ill patients with confirmed COVID-19.

DETAILED DESCRIPTION:
With the appearance of the COVID-19 pandemic, a race for the discovery of effective treatments to combat SARS-CoV-2 infection and its sequelae commenced. Some patients with COVID-19 develop severe acute respiratory syndrome which is the main reason for death. The aim of this study is to spearhead pharmacotherapeutic solutions for COVID-19 patients in the intensive care which have proven to be the hardest to treat due to the high death rate, the long-term allocation of patients in ICU, and the slow recovery that oftentimes leads to residual symptoms and signs. The ever-increasing pressure on the health care system requires finding an effective treatment that can benefit even advanced-stage patients such as those in the intensive care unit.

It was not until recently that the published literature about hydrogen sulfide shifted from revolving around its toxicity to its recognition as an endogenous gaseous signaling molecule and its biological roles. Hydrogen Sulfide (H2S) is a novel gaseous signaling molecule (gasotransmitter) that regulates a variety of physiological functions and provides protection against organ damage (anti-inflammatory, prolonged survival, cardioprotection, antioxidant, and more). H2S also displays beneficial roles in preventing lung disorders such as pneumonia, lung injury (acute/ chronic), and chronic obstructive pulmonary disease and limits viral replication. H2S has been shown to be effective in reversing lung inflammation and improving pulmonary function in various animal models. Based on preclinical data, cystathionine-γ-lyase (CSE)-derived H2S or exogenously applied H2S may block Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) entry into the host cells by interrupting Angiotensin-Converting Enzyme-2 (ACE2) and transmembrane protease serine-2 (TMPRSS2), inhibiting viral replication by attenuating syncytium formation and virus assembly/release, and thus may protect SARS-CoV-2-induced lung damage by suppressing the immune response and the development of inflammation.

Lymphopenia is a key characteristic of COVID-19 patients. Serum H2S was positively correlated with the lymphocyte count and is considered a predictor of mortality. Additionally reduced H2S bioavailability has been suggested as an indicator of enhanced pro-inflammatory responses and endothelial dysfunction. Both these conditions often accompany severe COVID-19. Interleukin-6 (IL-6) has been proposed as the principle pro-inflammatory cytokine involved in the cytokine storm that leads to severe lung injury, respiratory failure, and death by COVID-19. A negative association between IL-6 and serum H2S has been shown to exist. The above-mentioned results led to further evaluation of admission H2S levels as a marker of survival in a recent study. Results showed that serum levels of H2S on day 1 lower than 150.44 micromolars (μM) had the best tradeoff for sensitivity and specificity for death. Thus, administration of a H2S-donor could be a potential remedy for COVID-19 by relieving the damage in lungs and other organs.

Sodium thiosulfate (STS) is a H2S-donor with known safety and efficacy profile in humans for other diseases, including calciphylaxis and cyanide poisoning. STS can be metabolized to H2S and acts as a precursor for H2S signaling. Moreover, in patients presenting with acute coronary syndrome, a phase 1 study was conducted, showing that STS was well tolerated, even with concomitant use of blood pressure lowering drugs. Additionally, the Groningen Intervention study for Preservation of cardiac function with Sodium thiosulfate in ST-elevation myocardial infarction (GIPS-IV trial) is the first trial in humans designed to test the hypothesis that STS provides protection against I/R injury in patients presenting with ST-segment elevation myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or older than 18 years
2. Both genders
3. For women of childbearing potential, they must use or be willing to use a dual contraceptive method during the study.
4. Written consent statement provided by the patient or his / her legal representative in case patients are unable to consent.
5. Confirmed COVID-19 disease
6. WHO-CPS 7 to 9
7. Hospitalization in Intensive Care Unit
8. Serum H2S levels less than 140 μM

Exclusion Criteria:

1. Age less than 18 years
2. Denial of written consent
3. Decision not to resuscitate

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of treatment-emergent serious and non-serious adverse events between treatment groups. | Visit study day 28
  Change in the number of adverse events (AEs) and serious adverse events (SAEs) among treatment groups

SECONDARY OUTCOMES:
World Health Organization clinical progression scale (WHO-CPS) on day 7 from inclusion in the study | Visit study day 7
  Change in the WHO-CPS score on day 7 from inclusion in the study. The minimum WHO-CPS score is 0 for uninfected patients (no viral RNA detected) and the maximum is 10 for patients who are dead. Higher scores equals worse outcome
WHO-CPS on day 14 from inclusion in the study | Visit study day 14
  Change in the WHO-CPS score on day 14 from inclusion in the study. The minimum WHO-CPS score is 0 for uninfected patients (no viral RNA detected) and the maximum is 10 for patients who are dead. Higher scores equals worse outcome
WHO-CPS on day 28 from inclusion in the study | Visit study day 28
  Change in the WHO-CPS score on day 28 from inclusion in the study. The minimum WHO-CPS score is 0 for uninfected patients (no viral RNA detected) and the maximum is 10 for patients who are dead. Higher scores equal worse outcome
Average value of the total sequential organ failure assessment (SOFA) score on day 7 | Visit study day 7
  change between baseline sequential organ failure assessment (SOFA) score and measured sequential organ failure assessment SOFA score at Study Day 7. The minimum score is 0 points if the patient has PaO2/FiO2 (fraction of inspired oxygen) ≥400 mmHg, ≥150 Platelets (per mm3), hypotension (MAP ≥ 70mmHg), 15 on the Glasgow Scale, <1.2 bilirubin and creatinine or urine output (mg/dl). Maximum SOFA score is 24. if the patient has PaO2/FiO2 <100 mmHg, <20 Platelets (per mm3), Adrenaline >0.1 or Noradrenaline >0.1μg/kg/min , <6 on the Glasgow Scale, ≥12 bilirubin and ≥5.0 or <200ml/day creatinine or urine output (mg/dl).
Hydrogen sulfide concentrations daily until day 7 in patient's blood serum. | Visit study day 1 until visit day 7
  Change in patients blood serum concentrations of hydrogen sulfide levels from day 1 until day 7.
IL-6 cytokine concentrations daily until day 7 in patient's blood serum. | Visit study day 1 until visit day 7
  Change in patients blood serum concentrations of cytokine IL-6 levels from visit study day 1 until visit study day 7
Tumor Necrosis Factor (TNF) cytokine concentrations daily until day 7 in patient's blood serum. | Visit study day 1 until visit day 7
  Change in patients blood serum concentrations of cytokine TNF levels from visit study day 1 until visit study day 7
Change in the production of Th1, Th2, and T17 cytokines from mononuclear cells of patient's blood on days 1,4 and 7 | Visit study day 1, Visit study day 4, Visit study day 7
  Comparison of cytokine production on patients' blood serum by stimulation of monocytes, Th1, Th2, and T17 cells on visit study day 1, visit study day 4, and visit study day 7.
Ferritin concentrations on days 1,4 and 7 | Visit study day 1, Visit study day 4, Visit study day 7
  Changes in patients blood serum concentrations of ferritin levels on visit study day 1, visit study day 4 and visit study day 7
C-reactive protein concentrations on days 1,4 and 7 | Visit study day 1, Visit study day 4, Visit study day 7
  Changes in patients blood serum concentrations of C-reactive protein levels on visit study day 1, visit study day 4 and visit study day 7
D-dimers concentrations on days 1,4 and 7 | Visit study day 1, Visit study day 4, Visit study day 7
  Changes in patients blood serum concentrations of d-dimers levels on visit study day 1, visit study day 4 and visit study day 7
Cytokine IL-6 concentrations on days 1,4 and 7 | Visit study day 1, Visit study day 4, Visit study day 7
  Changes in patients blood serum concentrations of IL-6 levels on visit study day 1, visit study day 4 and visit study day 7

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Alamanos, MD, Principal Investigator — General Hospital of Athens KAT
Locations (1):
- General Hospitan of Athens KAT 2nd Department of ICU, Athens, Kifisia, Greece

IPD SHARING:
Plan to Share IPD: No